CLINICAL TRIAL: NCT06184776
Title: 'Lumbar Stiffness Disability Index' Turkish Adaptation, Reliability and Validity Study
Brief Title: 'Lumbar Stiffness Disability Index' Turkish Adaptation
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Elif Elcin Dereli, Professor, Istanbul Bilgi University
Other Study IDs: IstanbulBU1
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Adaptation; Lumbar Stiffness
Keywords: Adaptation; Reliability; Validity; Assessment; Lumbar Stiffness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Lumbar Stiffness Disability Index — The development and evaluation of the Turkish version of the Lumbar Stiffness Disability Index (LSDI) are planned. After ensuring the eligibility of adult participants included in the study, language validity will be established for the Turkish version of LSDI, and internal consistency will be assessed using Cronbach's alpha coefficient. Additionally, the test-retest reliability of the index will be evaluated by reapplying it to participants with a one-week interval. For external structure validity, LSDI scores will be correlated with Oswestry Disability Index, Functional Reach Test, and goniometric measurements. The study will include demographic data and measurements to examine the eligibility of individuals with specific medical conditions for the intervention.
  Other Names: Oswestry Disability Index; Functional Reach Test; Goniometric Measurements of Lumbar Region; Trunk Flexion and Hamstring Length Flexibility Test; Trunk Lateral Flexion Flexibility Test

SUMMARY:
Despite advancements in assessment and treatment methods, diagnosing and treating lower back pain remains challenging for researchers and clinicians. The literature doesn't support a definitive cause for the onset of back pain, as risk factors are diverse, population-specific, and inadequate when solely associated with back pain. Evaluating spinal stiffness is crucial, as it can either cause or result from back pain. However, assessing spinal stiffness lacks standardized and reliable methods, and studies regarding its relation to pain and movement are insufficient.

The measurement principles and optimization techniques for assessing spinal stiffness haven't been fully explained or practically recommended. Creating a practical diagnostic process involving examination procedures, a diagnostic checklist, and practical indices for evidence in clinical assessments is crucial. Early identification of individuals at risk of prolonged disability and illness is vital since specific interventions can be developed in the early stages.

The Lumbar Stiffness Disability Index (LSDI) stands out among valid and reliable tools for assessing lumbar stiffness and disability. It is an index designed in English, translated into languages like Chinese and Japanese, proving to be a useful tool to describe a patient's condition based on pain, function, and disability, tracking changes throughout treatment.

DETAILED DESCRIPTION:
Back pain is typically described as localized stiffness, often associated with muscle tension or in the lower border of the ribs and upper gluteal region, radiating or non-radiating to the leg. Back pain can be acute, subacute, or chronic, classified as such if it lasts less than six weeks, between six weeks and three months, or more than three months, respectively. Chronic back pain, especially, exhibits a high prevalence and continues to rise with industrialization, peaking in the 50-55 age group, with a notable increase in prevalence after the age of 80. It is more common in women. According to 2020 data from the World Health Organization, back pain has affected 619 million people globally, with an estimated increase to 843 million by 2050 due to population growth and aging. Back pain affects individuals of all age groups and is a leading cause of disability worldwide, imposing a significant financial burden on patients. Non-specific back pain accounts for approximately 90% of all cases.

Non-specific back pain poses a significant public health issue, lacking a sufficiently reliable and valid classification system for diagnosis in the literature. Imaging methods have limited effectiveness in diagnosis, as individuals with chronic back pain often present non-specific findings in imaging studies. Even asymptomatic patients frequently exhibit abnormal findings. Despite advancements in assessment and treatment methods, diagnosing and treating back pain remains challenging for both researchers and clinicians. The literature does not support a specific cause for the onset of back pain, as risk factors are diverse, population-specific, and associating back pain alone is inadequate.

Spinal segmental stiffness can either cause or result from back pain and is widely assessed in clinical and research settings. Despite frequent use of manual techniques in clinical assessments, the reliability of spinal stiffness assessment is weak, and studies on its relationship with pain and movement are insufficient. Existing reviews have not fully explained the principles of measurement methods for spinal stiffness or provided practical recommendations for optimizing measurements. To demonstrate evidence in clinical assessments, a practical diagnostic process involving examination procedures and a diagnostic checklist with a specific index is crucial. Early identification of individuals at risk of prolonged disability and illness is essential, as specific interventions can be developed in the early stages. Improvement becomes more challenging as symptoms persist and the condition becomes chronic.

When examining the literature, the Lumbar Stiffness Disability Index (LSDI) stands out among valid and reliable assessment tools for evaluating lumbar stiffness. Developed in English, translated into languages such as Chinese and Japanese, the LSDI is becoming widely recognized as a useful index for assessing lumbar spine rigidity and flexibility. The creation of a Turkish version of this index is considered valuable for clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals whose native language is Turkish,
* Those who are literate,
* Who have signed the voluntary consent form, and
* Who have been experiencing non-specific lower back pain for at least 3 months

Exclusion Criteria:

* Participants who are pregnant,
* Those who have experienced acute trauma related to the lumbar region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who has non-specific low back pain
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Lumbar Stiffness Disability Index | Baseline
  'Lumbar Stiffness Disability Index,' was developed by Hart et al. in 2013. It comprises 10 items and aims to assess the degree of impairment in the performance of daily activities due to the lack of mobility in individuals with compromised or lost lumbar spine flexibility. It queries the degree of execution of 10 movements related to the lumbar region in daily life, scored between 0 and 40, where a higher score indicates a higher level of disability (loss of ability). It can also be converted into a 100-point version. Developed as a 5-point Likert scale, it ranges from 0, indicating no impact and the activity being entirely achievable, to 4, meaning the activity is almost impossible to perform. Participants are asked to mark the value that is suitable for them in each activity.

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline
  The Oswestry Disability Index measures daily life activities from 10 different perspectives, including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual activity, social life, travel, and the varying degrees of pain. Each section contains 6 questions, and each question is scored between 0 and 5. The total score ranges from 0 to 50 and can be scaled to 100. This form is the most commonly used questionnaire for assessing disability due to back pain. Its validity and reliability have been demonstrated in the Turkish population, with a reported high level of internal consistency.
Functional Reach Test | Baseline
  It is used to assess the flexibility of the lumbar region while the participant is standing. The participant stands sideways to the wall, with the arm on the wall without touching it, shoulder in 90 degrees of flexion, elbow in extension, and the hand clenched into a fist. Meanwhile, the 3rd metacarpal head is placed against the wall at shoulder height, and the participant is expected to reach as far as possible. The changing 3rd metacarpal head is measured with a ruler. The distance between the starting and ending positions is calculated to obtain a score. Care should be taken to ensure that the participant's heels do not lift off the ground during forward bending. A reaching distance between 15-18 cm indicates limited functional balance, while a reaching distance of 25 cm and above indicates sufficient balance capacity. The testing will be repeated three times, and the average of the last two assessments will be used. 15-second breaks will be given between each repetition.
Goniometric Measurements of Lumbar Region | Baseline
  Goniometric measurements will be performed with a 360ᵒ universal goniometer. To ensure the smoothness of the measurement, the joint movement will be demonstrated to the participant beforehand. During the measurement, attention will be paid to the position of the pivot point, the moving arm, and the fixed arm. In the measurement of flexion and extension of the trunk, the lateral projection of the lumbosacral joint will be taken as the pivot point, and the fixed arm will be kept perpendicular to the ground, while the moving arm will follow the axillary midline. For the measurement of right and left lateral flexion, the 1st sacral spinous process will be considered as the pivot point, and the fixed arm will be kept perpendicular to the ground, while the moving arm will follow parallel to the 7th cervical spinous process.
Trunk Flexion and Hamstring Length Flexibility Test | Baseline
  The participant stands on a 15 cm block. They attempt to bend forward and touch their toes without bending their knees. The distance between the fingertip (distal end of the 3rd phalanx) and the block is measured. A positive value is recorded if it is below the block, and a negative value is recorded if it is above the block.
Trunk Lateral Flexion Flexibility Test | Baseline
  The participant stands with feet shoulder-width apart, arms by their side, in a standing position. The distal end of the 3rd phalanx of the hands is marked on the thigh. Subsequently, while flexing the trunk to the side (without leaning forward or backward), they are asked to slide their hand on the thigh. The point reached is marked, and the distance between the starting position and the marked point is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided